CLINICAL TRIAL: NCT05453214
Title: Safety and Efficacy of Fludrocortisone Addition to Dexamethasone in the Management of Hospitalised COVID-19 Patients
Brief Title: Mineralocorticoid Use in COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R111c/2021
Record Dates: First submitted 2022-07-09; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; ARDS
Keywords: fludrocortisone; mineralocorticoid; COVID-19; ARDS; Aldosterone
MeSH Terms: conditions — COVID-19 | interventions — fludrocortisone acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fludrocortisone arm (Experimental): 10 hospitalised COVID-19 patients meeting inclusion criteria will receive fludrocortisone 0.1 mg tablets in addition to dexamethasone 6 mg / 24 hours and standard care
  Interventions: Drug: Fludrocortisone Acetate 0.1 MG

INTERVENTIONS:
Drug: Fludrocortisone Acetate 0.1 MG — Fludrocortisone acetate 0.1 mg tablet / 12 hours; dose to be titrated according to response.

SUMMARY:
There is a considerable variability in aldosterone levels between individuals, and this may explain the wide variability in disease severity among those infected so we designed a pilot study to test for the safety and efficacy of fludrocortisone addition to standard of care in hospitalised COVID-19 patients.

DETAILED DESCRIPTION:
Many studies have shown involvement of renin-angiotensin-aldosterone system (RAAS) in pathophysiology of COVID-19. There is a considerable variability between people infected with SARS-COV-2 virus in terms of severity. At pathophysiological level there are variable degrees of increased capillary permeability with resultant fluid leak. We hypothesize that the physiological response to overcome this fluid leak mainly involves stimulation of mineralocorticoid (aldosterone) pathway. Hence; those with defective mineralocorticoid response are at high risk for disease complications.

Aldosterone secretion capacity is affected by many factors whether physiological (age, sex, ethnicity and pregnancy) or pathological (e.g. smoking); this is reflected in wide differences (regarding aldosterone levels) between groups of people depending on these factors.

These variations in mineralocorticoid capacity between groups of people may explain why some certain groups are at high risk for severe disease while others are at a lower risk.

So we designed this pilot study to assess safety and efficacy of mineralocorticoid, in the form of fludrocortisone, as a potential treatment for COVID-19 by its addition to dexamethasone in hospitalized COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female patients 18 years of age or older
* Diagnosed with COVID-19 pneumonia as per local guidelines
* Oxygen saturation (SaO2) of 93 % or less while they were breathing ambient air.

Exclusion Criteria:

* A physician decision that involvement in the trial will not be in the patient's best interest, presence of any condition that would not allow the protocol to be followed safely.
* known allergy or hypersensitivity to fludrocortisone.
* known severe liver or kidney disease, uncontrolled hypertension, diabetes mellitus and peptic ulcer disease.
* Hypokalemia (serum potassium of less than 3.5 mEq/L)
* Use of medications that are contraindicated with fludrocortisone and that could not be replaced or stopped during the trial period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-04 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Time to recovery | 28 days
  The first day, during the 28 days after enrollment, on which a patient met the criteria for category 1 or 2 on the eight-category ordinal scale

SECONDARY OUTCOMES:
Mortality Rate | 28 days
  All-cause mortality rate over 28 days post enrollment.
Length of hospital stay | 28 days
  Number of days since enrollment till hospital discharge.
Rate of ICU admission | 28 days
  Number of patients who experienced worsening of clinical status necessitating ICU admission.
Mechanical ventilation need | 28 days
  Number of patients who needed invasive mechanical ventilation during hospitalisation.
Improvement of lymphopenia | 7 days
  Reversal of lymphopenia - measured at days 3 and 7 after initiation of treatment.
Duration of Increased Supplemental Oxygen | 28 days
  Number of days counted from enrollment over which the participant requires supplemental oxygen in excess over his/her baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad S Zeafan, Principal Investigator — Alazhar allergy and immunology center
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in COVID-19. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after article publication and the data will be made accessible for up to 24 months
Access Criteria: Access to trial IPD can be requested by qualified researchers, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact muhammadsaberz@gmail.com

REFERENCES:
- [Background] Coto E, Avanzas P, Gomez J. The Renin-Angiotensin-Aldosterone System and Coronavirus Disease 2019. Eur Cardiol. 2021 Mar 9;16:e07. doi: 10.15420/ecr.2020.30. eCollection 2021 Feb. PMID 33737961
- [Background] Bauer JH. Age-related changes in the renin-aldosterone system. Physiological effects and clinical implications. Drugs Aging. 1993 May-Jun;3(3):238-45. doi: 10.2165/00002512-199303030-00005. PMID 8324299
- [Background] Wang W, Tang J, Wei F. Updated understanding of the outbreak of 2019 novel coronavirus (2019-nCoV) in Wuhan, China. J Med Virol. 2020 Apr;92(4):441-447. doi: 10.1002/jmv.25689. Epub 2020 Feb 12. PMID 31994742
- [Background] Szymanski P, Klisiewicz A, Lubiszewska B, Lipczynska M, Kowalski M, Janas J, Hoffman P. Gender differences in angiotensin II and aldosterone secretion in patients with pressure overloaded systemic right ventricles are similar to those observed in systemic arterial hypertension. Int J Cardiol. 2011 Mar 17;147(3):366-70. doi: 10.1016/j.ijcard.2009.09.535. Epub 2009 Nov 7. PMID 19896738
- [Background] Gossain VV, Sherma NK, Srivastava L, Michelakis AM, Rovner DR. Hormonal effects of smoking--I: Effects on plasma renin activity. Am J Med Sci. 1986 May;291(5):321-4. doi: 10.1097/00000441-198605000-00006. PMID 3518450